CLINICAL TRIAL: NCT06021470
Title: The StrokeCog Study: a Randomised Pilot Study of a Novel Cognitive Rehabilitation Intervention in Stroke
Brief Title: The StrokeCog Study: Cognitive Rehabilitation Intervention in Stroke
Acronym: StrokeCog-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StrokeCog-R
Record Dates: First submitted 2023-07-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-07

CONDITIONS: Stroke; Stroke Sequelae; Cognitive Impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Research Fellow conducting neuropsychological assessments will be blinded to random allocation and will not be involved in delivering the intervention. The neuropsychologist clinician will deliver the intervention and will not be involved in assessment or data analysis. The objective measures of cognition collected during the neuropsychological assessments are less subject to response bias than subjective assessments as patients cannot be blinded to treatment allocation; at post-assessment, patients will be asked not to reveal whether they have received the intervention or not in order to maximise researcher blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive rehabilitation intervention arm (Experimental): Five-week group-based and largely interactive format, with groups of four patients. Short presentations are delivered by the clinical neuropsychologist relating to psychoeducation and adjustment to stroke-related deficits in executive function, attention, and memory, respectively, and strategies addressing the activities and participation levels of functioning. Each session lasts approximately 2.5 hours, with a break in the middle. Tailored home activities are included for completion between group sessions to encourage self-efficacy and generalisation of skills and strategies. A member of the research team contacts all participants by telephone twice a week to assess engagement and reported self-efficacy in managing cognitive difficulties. In addition, a weekly text message is sent to all participants. In the proposed pilot RCT, for those receiving the intervention, the text message will contain tips on implementing compensatory strategies.
  Interventions: Behavioral: Cognitive rehabilitation intervention
- Usual care (No Intervention): Those in the control group will be allocated to usual care from their multidisciplinary rehabilitation team in both acute and rehabilitation settings. Usual rehabilitation care is likely to vary across hospital settings (acute vs. rehabilitation). Information about type, dose, and amount of rehabilitation therapy will be captured from patients' medical charts in both the intervention and control arm of the study.
  A member of the research team (RA) contacts all participants by telephone twice a week to assess engagement and reported self-efficacy in managing cognitive difficulties. In addition, a weekly text message is sent to all participants. For those in the wait-list control condition, the text message will contain a positive affirmation.

INTERVENTIONS:
Behavioral: Cognitive rehabilitation intervention — The intervention comprises a five-week group-based cognitive rehabilitation intervention delivered by a clinical neuropsychologist, with home activities tailored to each stroke survivor's identified goals. Sessions involve four patients and are delivered once per week lasting 2.5 hours with breaks.
  Arms: Cognitive rehabilitation intervention arm

SUMMARY:
This study aims to progress to the next stage of feasibility testing, by conducting a pilot randomised controlled study with consecutive stroke patients who have mild to moderate cognitive impairment following stroke. The primary focus of the proposed randomised pilot RCT is on recruitment and retention of patients in the intervention, and follow-up assessments. The researchers will also investigate outcomes associated with the intervention and the anticipated effect size for powering a larger trial, with a focus on the feasibility of implementing the intervention in a future definitive randomised controlled trial. The researchers will also carry out a study within a trial (SWAT), comparing recruitment and retention rates across acute, rehabilitation and chronic stroke settings.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability in Ireland and worldwide. Many people are aware of the physical disabilities that occur following stroke, but are less aware of the cognitive problems that people experience. Cognitive problems, or cognitive impairment, include difficulties with thinking, memory and concentration. They affect up to 60% of people after stroke. Stroke survivors and their families describe cognitive impairment as one of the most difficult stroke outcomes to deal with, and the biggest obstacle to returning to pre-stroke life.

Rehabilitation of post-stroke cognitive impairment has received little attention compared with physical rehabilitation. Current evidence indicates that cognitive impairment continues to decline and - especially if the person has another stroke - develops into dementia, one of the main reasons people move to long-term, or nursing home, care (LTC). Intervening to rehabilitate cognitive impairment may halt further decline and/or improve cognitive function, thus improving quality of life, and preventing progression to dementia and LTC.

The StrokeCog research team has developed a cognitive intervention based on extensive review of international studies and in-depth consultation with people who have had a stroke, their family members, and healthcare professionals working with people following stroke. The researchers have already tested this intervention with a very small number of patients with stroke-related cognitive impairment. Working with patient representatives, this research programme seeks to further test this intervention with a larger sample of patients with stroke-related cognitive problems. The researchers will collect information on the best way to recruit patients into the study, how many complete the intervention, and examine initial results on the benefits of the intervention. The team will collect and analyse detailed information on the costs associated with delivering this intervention. The study will provide strong evidence on whether the intervention is worthy of further investigation in a larger-scale research trial.

ELIGIBILITY:
Inclusion Criteria:

1. WHO-defined stroke, to include ICD-10 codes 160 (subarachnoid haemorrhage), 161 (intracerebral haemorrhage), 163 (cerebral infarction) including sub-categories, and 164 (stroke not specified as haemorrhage or infarction);
2. First-ever and recurrent stroke;
3. Age 18 and over (no upper age limit);
4. Community dwelling (i.e., normal place of residence is not in a long-term care facility)
5. Is a resident in the Republic of Ireland
6. Capable of providing informed consent

Exclusion Criteria:

1. Transient ischaemic attack;
2. Aphasia;
3. Poor English language ability;
4. Nursing home resident;
5. Dementia or severe cognitive impairment;
6. Neurodegenerative disorder;
7. Current psychiatric disorder (as defined by DSM-V or ICD-II criteria);
8. Terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Digit Span forward & backward (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
Verbal Fluency (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
Colour Trails Tests A&B (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
15-Item modified Boston Naming Test (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
Symbol Digit Modalities Test (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
Rey Complex Figure Test copy, immediate/delayed recall, and recognition (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.
Hopkins Verbal Learning Test - immediate/delayed recall, & recognition (National Institute of Neurological Disorders & Stroke (NINDS) Assessment Battery) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The primary outcome is cognitive function, assessed using the standardised National Institute of Neurological Disorders & Stroke (NINDS) Assessment battery. The primary outcome will be used for purposes of estimating the effect size (including standard deviation) to inform a power calculation for estimation of sample size for a definitive trial.

SECONDARY OUTCOMES:
Goal Attainment Scaling based on SEIQoL (Self-efficacy in managing cognitive deficits) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Modified Stroke Self-Efficacy Scale (Self-efficacy in managing cognitive deficits) | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Test of Premorbid Functioning | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Wechsler Abbreviated Scale of Intelligence | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Fatigue Severity Scale | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
General Anxiety Disorder 7-item assessment | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Patient Health Questionnaire | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Modified Rankin Scale | Patients will complete these cognitive assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  A major secondary outcome is patient-reported self-efficacy in managing their cognitive deficits.
  Additionally, personal and demographic details will be recorded for each patient. Mood, functional ability, quality of life (QoL), adherence, and recurrent stroke will be assessed as important secondary outcome measures.
Patient Health Questionnaire (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.
General Anxiety Disorder 7-item assessment (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.
Vulnerable Elders Survey (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.
Zarit Burden Interview (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.
Perceived Stress Scale (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.
Informant Questionnaire for Cognitive Decline in the Elderly, short form (Family member/carer outcome) | Carers/family members will complete these assessments at three time points: prior to (1) and following (2) the 5-week group based rehabilitation period (or control period), and at four months post-intervention (3).
  The patient's family member/carer will be asked to complete a relative/carer assessment.

OTHER OUTCOMES:
Eligibility rates (Intervention feasibility) | Through study completion, an average of 1.5 years
  This study will provide robust evidence to inform a decision to progress to a definitive trial, including eligibility, recruitment, and retention rates, feasibility of randomisation, acceptability to patients, and resource use based on micro-costing of the intervention delivery.
Recruitment rates (Intervention feasibility) | Through study completion, an average of 1.5 years
  This study will provide robust evidence to inform a decision to progress to a definitive trial, including eligibility, recruitment, and retention rates, feasibility of randomisation, acceptability to patients, and resource use based on micro-costing of the intervention delivery.
Retention rates (Intervention feasibility) | Through study completion, an average of 1.5 years
  This study will provide robust evidence to inform a decision to progress to a definitive trial, including eligibility, recruitment, and retention rates, feasibility of randomisation, acceptability to patients, and resource use based on micro-costing of the intervention delivery.
Feasibility of Randomisation (Intervention feasibility) | Through study completion, an average of 1.5 years
  This study will provide robust evidence to inform a decision to progress to a definitive trial, including eligibility, recruitment, and retention rates, feasibility of randomisation, acceptability to patients, and resource use based on micro-costing of the intervention delivery.
Resource Use (Microcosting)(Intervention feasibility) | Through study completion, an average of 1.5 years
  Micro-costing of materials and consumables utilised in the pilot study and the staffing costs and time taken to recruit patients, and costs associated with the usual care comparator will be recorded
Qualitative Process Evaluation (Intervention Acceptability) | Through study completion, an average of 1.5 years
  Qualitative data will be separately collected from patients and staff involved in the intervention in the form of focus group interviews to explore how they experienced the intervention process and to indicate the extent to which it was found to be helpful and/or feasible.